CLINICAL TRIAL: NCT01481181
Title: An Efficacy Trial of a Gravity Fed Household Water Treatment Device as a Delivery System for Zinc in Zinc Deficient Children and Women From Low Income Settings
Brief Title: An Efficacy Trial of a Gravity Fed Household Water Treatment Device as a Delivery System for Zinc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LSF Zinc Kisumu study
Record Dates: First submitted 2011-11-11; First posted 2011-11-29 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Diarrhoea
Keywords: zinc water diarrhoea growth preschool children
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- zinc enriched water (Experimental): zinc enriched purified water at 2-6mg/l per day
  Interventions: Dietary Supplement: Zinc enriched water
- purified water only (No Intervention): non zinc enriched, purified drinking water
- control group (No Intervention): group of households receiving hygiene practice recommendations and water guard (water purifying solution)

INTERVENTIONS:
Dietary Supplement: Zinc enriched water — 3mg zinc/L of purified water from a filter installed in the households
  Arms: zinc enriched water

SUMMARY:
In low-income settings in developing countries unsafe water is one of the leading causes of high prevalence of waterborne diseases such as diarrhoea.Zinc is an essential trace element that has a critical role in growth and immunity. Supplementation with zinc is considered effective in reducing morbidity from diarrhoeal and other infectious diseases. Verstergaard Frandsen S.A. (Switzerland) has developed a point-of-use water filtration system called LifeStraw®Family (LSF) that removes water's turbidity, reduces the microbiological contamination and enriches water with zinc at a concentration of 3.5 mg/L. The objective of the study is to assess the efficacy of LSF to increase the zinc status (serum zinc concentration) and intake in Kenyan children aged 2-5years with zinc deficiency.The study hypotheses are:

A. Use of the LSF device will reduce microbiological contamination of the household supply of drinking and cooking water; B. Use of the LSF device will increase zinc intakes in preschool children; C. Use of the LSF device will increase serum zinc concentration in preschool children; D. Achieving A, B and C will improve growth in preschool children; E. Achieving A, B and C will reduce the frequency and duration of diarrheal disease in preschool children and in members of the participating households.

DETAILED DESCRIPTION:
Introduction: In low-income settings in developing countries unsafe water is one of the leading causes of high prevalence of waterborne diseases such as diarrhoea. Point-of-use water treatment systems are currently considered by UNICEF as more effective in delivering safe drinking water than interventions applied at source. Zinc is an essential trace element that has a critical role in growth and immunity. Supplementation with zinc is considered effective in reducing morbidity from diarrhoeal and other infectious diseases. Verstergaard Frandsen S.A. (Switzerland) has developed a point-of-use water filtration system called LifeStraw®Family (LSF) that removes water's turbidity, reduces the microbiological contamination and enriches water with zinc at a concentration of 3.5 mg/L.

Objective: To assess the efficacy of LSF to increase the zinc status (serum zinc concentration) and intake in Kenyan children aged 2-5years with zinc deficiency.

Study Design and Methods: A study population living in an area with low Zn status and sharing the same unimproved water supply will be included in the trial and randomly assigned to one of the treatment groups for 12 months. All households will receive hygiene practice recommendations (HPRs). In addition to HPR, group one will receive the LSF device with the zinc delivery system; group 2 will receive HPRs and a LSF without zinc delivery system, and group 3 will receive HPRs. At baseline, mid-point and end-point, anthropometrics (weight, height, mid-upper arm circumference MUAC), and 7 ml whole blood will be collected from preschool children for determination of SZn, C-reactive protein (CRP), hemoglobin (Hb) and serum ferritin (SF). Children and adult subjects remaining zinc deficient at completion of the trial will receive zinc supplements.

Expected outcome: This study will investigate the efficacy of a water treatment device as a means to provide Zn in communities where high prevalence of surface water use and zinc deficiency coexists. Increasing the microbiological quality of water and the contemporaneous low dose fortification with zinc, could prove useful in the global effort to control zinc deficiency and increase the supply of clean drinking water

ELIGIBILITY:
Inclusion Criteria:

* Children found to have serum zinc concentration <65μg/dL at pre screening.
* Women that have become pregnant during the study.

Exclusion Criteria for children:

* Subjects with severe anemia (Hb<7g/dl)
* Subjects with severe zinc deficiency (SZn<40 μg/dL)
* Subjects receiving zinc supplementation
* Subject with chronic diseases affecting zinc metabolism, such as kidney diseases or chronic gastrointestinal disease.
* Subjects participating in any other clinical trials in the study site

Exclusion criteria for women:

* Women not residing in the study area until childbirth
* Subjects with severe anemia (Hb<7g/dl)
* Subjects with sever zinc deficiency (SZn<40 μg/dL)
* Subjects receiving zinc supplementation
* Subject with chronic diseases affecting zinc metabolism, such as kidney diseases or chronic gastrointestinal disease.
* Subjects currently enrolled in other clinical trials in other trials on the study site

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 270 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
zinc status | one year
  At baseline, endpoint and at a randomly assigned screening between month 1 and 11, a 6 ml whole blood sample will be collected by venipuncture in 2-5y children (N=270). The blood sample will be used to determine concentration of zinc in the serum (SZn). Inflammation indicator C-reactive protein (CRP) will be analysed to adjust SZn values.

SECONDARY OUTCOMES:
rates of diarrhoea and growth in preschool children | one year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmerman, MD, PhD, Principal Investigator — ETH Zurich , Wageningen University; Diego Moretti, PhD, Principal Investigator — Wageningen University
Locations (1):
- Maseno University, School of Public health, Kisumu, Western Kenya, Kenya